CLINICAL TRIAL: NCT02541188
Title: Genotype and Phenotype in Early Onset Breast Cancer in Young Women on the Two Shores of the Mediterranean Sea
Acronym: MediSein
Status: Terminated | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF 9428
Record Dates: First submitted 2015-08-26; First posted 2015-09-04 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- breast cancer in young women is in the Maghreb: breast cancer in young women (< 40years old) is in the Maghreb
  Interventions: Genetic: Genetic analysis
- Breast cancer in young women in the western countries: Breast cancer in young women (< 40years old) in the western countries
  Interventions: Genetic: Genetic analysis

INTERVENTIONS:
Genetic: Genetic analysis

SUMMARY:
Breast cancer are common on mediterranean basin. Epidemiological data suggest that breast cancer in young women (< 40years old) is more aggressive in the Maghreb countries comparatively to western countries. This aggressiveness could be associated with phenotypic and genotypic differences between this two populations.

DETAILED DESCRIPTION:
The object of this study is to compare the genotypic and phenotypic differences between south and north shore of the mediterranean sea.

ELIGIBILITY:
Inclusion Criteria:

* Patient have or have had a breast cancer diagnosed before 40 years old
* Breast cancer proven by histology
* BRCA1/2 analysis proposed, realized, ongoing
* Women >18 years old
* Patient with insurance
* Patient informed and no-opposed

Exclusion Criteria:

* Patient have or have had a breast cancer diagnosed after 40 years old
* Patient requiring tutorship or guardianship
* Adult patient protected by law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients have or have had a breast cancer diagnosed before 40 years old in two shores of the Mediterranean sea (France, lgeria, Marocco, Egypt, Tunisia)
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2016-10-02 (Actual); Study Completion 2017-01-02 (Actual)

PRIMARY OUTCOMES:
Genetic analysis of Breast Cancer susceptibility gene 1 (BRCA 1) | The day of inclusion
Genetic analysis of Breast Cancer susceptibility gene 2 (BRCA 2) | The day of inclusion

SECONDARY OUTCOMES:
Analysis TNM grade | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)
Analysis histoprognostic grade Scarf Bloom and Richardson (SBR) | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)
analysis of hormone receptor ER | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)
growth factors analysis (Ki 67) | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)
analysis of HER2 | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)
analysis of hormone receptor PR | The day of inclusion
  Tumors will be phenotyped by giving the histological characteristics (TNM and SBR grade, hormone receptors (ER, PR), growth factors (Ki 67) and HER2)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PUJOL, MDPhD, Principal Investigator — Oncogenetic Unit -CHU de Montpellier
Locations (1):
- CHU de Montpellier, Montpellier, France